CLINICAL TRIAL: NCT00581464
Title: Healthier Hearts and Brains in Treating Smoking: The HABITS Study
Acronym: HABITS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO08030007
Record Dates: First submitted 2007-12-20; First posted 2007-12-27 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Smoking
Keywords: Smoking cessation; Tobacco dependence; Mindfulness; fMRI; Craving
MeSH Terms: conditions — Smoking; Smoking Cessation; Tobacco Use Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Behavioral: Standard Behavioral Therapy
- 2 (Active Comparator)
  Interventions: Behavioral: Mindfulness Based Addiction Therapy

INTERVENTIONS:
Behavioral: Standard Behavioral Therapy — Standard therapy to help participants with smoking cessation.
  Arms: 1
Behavioral: Mindfulness Based Addiction Therapy — A novel mind body therapy that extends basic behavioral therapy principles to include the practice of mindfulness, which fosters a dispassionate approach to the experience of craving.
  Arms: 2

SUMMARY:
80 nicotine dependent adults ages 18-65 who desire to quit smoking will be screened and, if eligible, enrolled and randomized to one of two four-week treatments for smoking cessation. The treatments are standard behavioral therapy and Mindfulness Based Addiction Therapy (MBAT), which is standard therapy plus mindfulness. Standard therapy and MBAT incorporate elements of widely-used tools for smoking cessation including managing craving and strong emotions, problem solving, tips on healthy eating and keeping active, and exercises based on cognitive and behavioral therapy. MBAT uniquely incorporates mindfulness practice (a relaxation therapy) into standard therapy. Participants complete questionnaires and undergo an fMRI scan at baseline and at the end of therapy (after they complete the 4 weeks of standard therapy or MBAT). During each scan, participants will complete a validated smoking-related cue paradigm and a validated affect labeling paradigm.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be considered eligible for enrollment if they are between 18-65 years old, smoke at least ½ pack cigarettes per day, desire to quit smoking (self-reported 75+ out of a possible 100), and have no contraindications for varenicline medication therapy or fMRI scanning (such as body weight over 250 lbs, intravascular metal devices including stents, or claustrophobia).

Exclusion Criteria:

* Participants will not be considered eligible for enrollment if they are not between 18-65 years old, smoke less than ½ pack cigarettes per day, do not desire to quit smoking (self-reported -75 out of a possible 100), or have contraindications for varenicline medication therapy or fMRI scanning (such as body weight over 250 lbs, intravascular metal devices including stents, or claustrophobia).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2009-11; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Smoking Cessation | week 2 and 6 month follow-up

SECONDARY OUTCOMES:
Exhaled CO readings | baseline, weeks 2-4, post class follow-up, long term follow-up
Saliva Test | baseline
Functional Magnetic Resonance Imaging | baseline & follow-up
Urine Pregnancy Test | baseline & follow-up
Nicotine Replacement Therapy | Week 1
Self Reported Measures | baseline, post class follow-up & long term follow-up
Standard Cognitive Therapy | weeks 1-4
Mindfulness Based Cognitive Therapy | weeks 1-4

CONTACTS AND LOCATIONS:
Overall Officials: Hilary Tindle, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States